CLINICAL TRIAL: NCT03265535
Title: Validation of a Single Rest-Stress Imaging Protocol for Myocardial Perfusion Imaging
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Georges El Fakhri, Director, Gordon Center for Medical Imaging, Massachusetts General Hospital
Other Study IDs: 2016P002531
Record Dates: First submitted 2017-08-25; First posted 2017-08-29 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Coronary Artery Disease; Myocardial Ischemia
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Healthy Volunteers: Subjects without history of coronary artery disease
  Interventions: Diagnostic Test: Single-Scan Two-Injection Protocol
- Subjects with coronary artery disease: Subjects with coronary artery disease and abnormal SPECT myocardial perfusion imaging within the last 12 months
  Interventions: Diagnostic Test: Single-Scan Two-Injection Protocol

INTERVENTIONS:
Diagnostic Test: Single-Scan Two-Injection Protocol — Single-Scan Two-Injection Protocol

SUMMARY:
We propose a single-scan two-injection myocardial perfusion imaging protocol using ammonia. Subjects will undergo single-scan two-injection imaging as well as regular stress single-scan single-injection protocol and the myocardial blood flow of both techniques will be compared.

ELIGIBILITY:
Healthy Volunteers:

Inclusion Criteria:

* Subjects must be ≥30 and ≤75 years of age;
* Subjects must provide informed consent prior to study procedures;

Exclusion Criteria:

* History of CAD, including:
* Prior abnormal myocardial perfusion study
* History of MI
* History of angina
* Coronary artery obstruction >50% on CTA and/or angiography
* Left ventricular ejection fraction <50%
* Any relative or absolute contraindication to adenosine stress, including:
* 2nd or 3rd degree heart block
* Bradycardia (HR<50 bpm)
* Recent acute coronary syndrome (ACS)
* Unstable angina
* Severe heart failure (left ventricular ejection fraction <15%)
* Ventricular arrhythmia
* Severe asthma and/or chronic obstructive pulmonary disease (COPD)
* Baseline hypotension defined as systolic blood pressure < 90 mmHg
* Caffeine intake within 24 hours prior to imaging
* Current use of theophylline, dipyridamole, or carbamazepine
* Allergy or intolerance to adenosine
* Positive serum and/or urine pregnancy test, or lactating, or possibility of pregnancy cannot be ruled out prior to dosing;

Subjects with CAD:

Inclusion criteria

* Subjects must be ≥30 and ≤75 years of age;
* Subjects must provide informed consent prior to study procedures;
* Abnormal myocardial perfusion study within the past 12 months

Exclusion criteria

* Revascularization (percutaneous coronary intervention and/or coronary artery bypass) following last myocardial perfusion study
* Acute coronary syndrome within 30 days
* Left ventricular ejection fraction <50%
* Any relative or absolute contraindication to adenosine stress, including:
* 2nd or 3rd degree heart block
* Bradycardia (HR<50 bpm)
* Recent acute coronary syndrome (ACS)
* Unstable angina
* Severe heart failure (left ventricular ejection fraction <15%)
* Ventricular arrhythmia
* Severe asthma and/or chronic obstructive pulmonary disease (COPD)
* Baseline hypotension defined as systolic blood pressure < 90 mmHg
* Caffeine intake within 24 hours prior to imaging
* Current use of theophylline, dipyridamole, or carbamazepine
* Allergy or intolerance to adenosine
* Any clinically significant acute or unstable physical or psychological disease, judged by the investigators, to be incompatible with the study;
* Radiation exposure exceeds current Radiology Department guidelines (i.e. 50 mSv in the prior 12 months);
* Female participants only: Positive serum and/or urine pregnancy test, or lactating, or possibility of pregnancy cannot be ruled out prior to dosing;
* Inability to provide written informed consent;

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients of the Massachusetts General Hospital
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-09-21 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Stress MBF | Single session (<2 hours)
  Difference in stress myocardial blood flow measured by the single-scan two-injection protocol versus conventional single-scan single-injection stress protocol

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No